CLINICAL TRIAL: NCT07105150
Title: Efficacy of an Educational Video-Based Program to Treat Urinary Incontinence in Women Referred for Pelvic Floor Rehabilitation
Brief Title: Efficacy of a Video-Based Educational Program on Female Urinary Incontinence
Acronym: EVRP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-A00419-40
Record Dates: First submitted 2025-07-12; First posted 2025-08-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinence; pelvic floor rehabilitation; video-based program; education
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- video-based education program group (Experimental)
  Interventions: Behavioral: video-based education program
- written information group (Active Comparator)
  Interventions: Other: written information

INTERVENTIONS:
Behavioral: video-based education program — The video-based education program will include 4 workshops of 20 minutes each, at a rate of 1 video per week:
  Video 1: Anatomy and physiology of the pelvic floor; Video 2: Physiology of the urinary tract; Video 3: Physiology of the digestive tract; Video 4: Pathophysiology of urinary incontinence and other pelvic floor disorders (genital prolapse and anal incontinence) and preventive measures in daily activities.
  Arms: video-based education program group
Other: written information — The control group will receive a paper information document (containing the same information as the intervention group) during the 4-week period
  Arms: written information group

SUMMARY:
The aim of this clinical trial is to assess the effectiveness of a 4-week video-based education program in enhancing urinary continence among women with urinary incontinence referred for pelvic floor rehabilitation

The main question it aims to answer is :

• Does a structured video-based education program reduce the symptoms of urinary incontinence before any pelvic floor muscle strengthening ? Researchers will compare this program to a paper document (providing similar information) to see if this improves urinary continence in women suffering from urinary incontinence.

Participants will :

* receive either the video-based education program or a paper information document (providing similar information) prior to the sessions with the physiotherapist
* then follow pelvic floor rehabilitation sessions with the physiotherapist according to usual practice
* complete the urinary incontinence questionnaire after the 4-week video education program (intervention group) or 4 weeks after receiving the paper document (control group), and after each pelvic floor rehabilitation session with the physiotherapist and at the end of the sessions
* will be monitored at 1 and 2 years to evaluate urinary incontinence following the intervention.

DETAILED DESCRIPTION:
The video-based education program will include 4 workshops of 20 minutes each, at a rate of 1 video per week:

Video 1: Anatomy and physiology of the pelvic floor; Video 2: Physiology of the urinary tract; Video 3: Physiology of the digestive tract; Video 4: Pathophysiology of urinary incontinence and other pelvic floor disorders (genital prolapse and anal incontinence) and preventive measures in daily activities.

ELIGIBILITY:
Inclusion Criteria:

* Any woman referred for pelvic floor rehabilitation sessions for urinary incontinence (defined as 'any involuntary leakage reported by the patient' according to the International Continence Society)
* Women requiring perineal rehabilitation for urinary incontinence
* Aged 18 years or older
* Having access to a connected device (tablet, smartphone, computer)
* Having a functional email address
* Covered by a social security scheme
* Informed, and written consent (signed by the participant and the investigator)

Exclusion Criteria:

* Women unable to complete questionnaires (unable to read French or unable to write)
* Visually impaired individuals who cannot watch the video or read the printed material
* Genital prolapse extending beyond the hymen
* Documented neurological disorders
* Individuals receiving psychiatric care and those unable to express their consent
* History of pelvic fractures or dorsolumbar surgery
* Chronic pelvic pain
* Women who have given birth within the last 6 month
* Individuals with enhanced protection: minors, individuals deprived of liberty, individuals residing in a health or social institution, pregnant or breastfeeding women, adults under legal protection, and patients in emergency situations.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2026-01-09 (Actual); Primary Completion 2028-02-15 (Estimated); Study Completion 2030-01-09 (Estimated)

PRIMARY OUTCOMES:
Urinary incontinence score comparison between the 2 groups | At the end of the video-based education program (5 weeks after inclusion)
  the urinary incontinence score will measured using the ICIQ-SF (International Consultation on Incontinence Questionnaire-Short Form), ranging from 0 (corresponding to 'no urinary incontinence') to 21 (corresponding to 'very severe urinary incontinence'), collected after the video-based education program in the intervention group (scheduled over 4 weeks) and within the same timeframe in the control group (which received only the information document)

SECONDARY OUTCOMES:
Urinary incontinence score evolution in the intervention group | from inclusion until the end of the video education program (5 weeks after inclusion)
  Change in urinary incontinence score (International Consultation on Incontinence Questionnaire- Short Form, ICIQ-SF, ranging from 0 = 'no incontinence' to 21 = 'very severe incontinence') between inclusion and the end of the video education program in the intervention group (scheduled over 4 weeks)
Urinary incontinence score evolution in the control group | from inclusion to 5 weeks following the distribution of the paper information document
  Change in urinary incontinence score (International Consultation on Incontinence Questionnaire- Short Form, ICIQ-SF, ranging from 0 = 'no incontinence' to 21 = 'very severe incontinence') between inclusion and 5 weeks following the distribution of the paper information document
Number of pelvic floor rehabilitation sessions required in the intervention group | ICIQ-SF score recorded after each pelvic floor rehabilitation session, through end of rehabilitation, an average of 3 months
  The number of rehabilitation sessions needed to achieve a reduction of 3 points or more in the urinary incontinence score (ICIQ-SF) - a difference considered clinically significant - or a reduction of less than 3 points, provided that the decrease is deemed sufficient or satisfactory by the physiotherapist
Number of pelvic floor rehabilitation sessions required in the control group | ICIQ-SF score recorded after each pelvic floor rehabilitation session, through end of rehabilitation, an average of 3 months
  The number of rehabilitation sessions needed to achieve a reduction of 3 points or more in the urinary incontinence score (ICIQ-SF) - a difference considered clinically significant - or a reduction of less than 3 points, provided that the decrease is deemed sufficient or satisfactory by the physiotherapist
Urinary incontinence score evolution during the pelvic floor rehabilitation sessions in the intervention group | ICIQ-SF score recorded after each pelvic floor rehabilitation session, through end of rehabilitation, an average of 3 months
  The variation in the urinary incontinence score (ICIQ-SF) from first pelvic floor rehabilitation session to the 10th session and up to the last session
Urinary incontinence score evolution during the pelvic floor rehabilitation sessions in the control group | ICIQ-SF score recorded after each pelvic floor rehabilitation sessions, through end of rehabilitation, an average of 3 months
  The variation in the urinary incontinence score (ICIQ-SF) from first pelvic floor rehabilitation session to the 10th session and up to the last session
Quality of life score evolution in the intervention group | at inclusion and after the video-based education program (5 weeks after inclusion) , as well as between inclusion and at the end of the pelvic floor rehabilitation sessions, an average of 3 months
  The difference in the quality of life score associated with urinary symptoms (specific CONTILIFE questionnaire) and general quality of life (EuroQoL-5D questionnaire) at inclusion and after the video-based education program , as well as between inclusion and at the end of the pelvic floor rehabilitation sessions
Quality of life score evolution in the control group | at inclusion and 5 weeks after the distribution of the paper document information, as well as between inclusion and at the end of the pelvic floor rehabilitation sessions, an average of 3 months
  The difference in the quality of life score associated with urinary symptoms (specific CONTILIFE questionnaire) and general quality of life (EuroQoL-5D questionnaire) at inclusion and 5 weeks after the distribution of the paper document information, as well as between inclusion and at the end of the pelvic floor rehabilitation sessions
Pelvic floor and sexual symptoms scores evolution in the intervention group | between inclusion and the end of the video-based education program (5 weeks after inclusion), as well as between inclusion and the end of the pelvic floor rehabilitation sessions, an average of 3 months
  The difference in the score for pelvic floor and sexual symptoms that may be associated with urinary incontinence (FPFQ - Female Pelvic Floor Questionnaire) between inclusion and the end of the video-based education program, as well as between inclusion and the end of the pelvic floor rehabilitation sessions
Pelvic floor and sexual symptoms scores evolution in the control group | at inclusion and 5 weeks after the distribution of the paper information document, as well as between inclusion and the end of the pelvic floor rehabilitation sessions, an average of 3 months
  The difference in the score for pelvic floor and sexual symptoms that may be associated with urinary incontinence (FPFQ - Female Pelvic Floor Questionnaire) between inclusion and 4 weeks after the distribution of the paper information document, as well as between inclusion and the end of the pelvic floor rehabilitation sessions
Patient-perceived improvement score evolution in the intervention group | after the video-based education program (5 weeks after inclusion)and at the end of the pelvic floor rehabilitation sessions, an average of 3 months
  Patient-perceived improvement score evaluated by the PGII (Patient Global Impression of Improvement) questionnaire after the video-based education program and at the end of the pelvic floor rehabilitation sessions
Patient-perceived improvement score evolution in the control group | 5 weeks after inclusion and at the end of the pelvic floor rehabilitation sessions, an average of 3 months
  Patient-perceived improvement score evaluated by the PGII (Patient Global Impression of Improvement) questionnaire 5 weeks after the distribution of the paper information document and at the end of the pelvic floor rehabilitation sessions
Patient-perceived improvement score evolution according to the urinary incontinence type in the intervention group | after the video-based education program (5 weeks after inclusion) and at the end of the pelvic floor rehabilitation sessions, an average of 3 months)
  Patient-perceived improvement score evaluated by the PGII (Patient Global Impression of Improvement) questionnaire after the video-based education program and at the end of the pelvic floor rehabilitation sessions, according to the urinary incontinence type (Stress urinary incontinence, Urge urinary incontinence and mixed incontinence)
Patient-perceived improvement score evolution according to the type of urinary incontinence | 5 weeks after inclusion and at the end of the pelvic floor rehabilitation sessions, an average of 3 months
  Patient-perceived improvement score evaluated by the PGII (Patient Global Impression of Improvement) questionnaire 5 weeks after the distribution of the paper information document and at the end of the pelvic floor rehabilitation sessions, according to the urinary incontinence type (Stress urinary incontinence, Urge urinary incontinence and mixed incontinence)
Patient-perceived improvement score evolution according to the dimensions of the Urinary Leakage Circumstances questionnaire in the intervention group | after the video-based education program (5 weeks after inclusion) and at the end of the pelvic floor rehabilitation sessions, an average of 3 months
  Patient-perceived improvement score evaluated by the PGII (Patient Global Impression of Improvement) questionnaire after the video-based education program and at the end of the pelvic floor rehabilitation sessions, according to the dimensions of the Urinary Leakage Circumstances questionnaire (ULCQ)
Patient-perceived improvement score evolution according to the dimensions of the Urinary Leakage Circumstances questionnaire in the control group | 5 weeks after inclusion and at the end of the pelvic floor rehabilitation sessions, an average of 3 months
  Patient-perceived improvement score evaluated by the PGII (Patient Global Impression of Improvement) questionnaire 5 weeks after the disctribution of the paper information document and at the end of the pelvic floor rehabilitation sessions, according to the dimensions of the Urinary Leakage Circumstances questionnaire (ULCQ)
ICIQ-SF score evolution 12 and 24 month after the end of the pelvic floor rehabilitation sessions in the intervention group | at the end of the pelvic floor rehablitation sessions and after 12 and 24 months
  Difference between the ICIQ-SF score at the end of the pelvic floor rehablitation sessions and the ICIQ-SF score at 12 months and at 24 months in the intervention group
ICIQ-SF score evolution at 12 and 24 months after the end of the pelvic floor rehabilitation sessions | at the end of the pelvic floor rehablitation sessions and after 12 and 24 months
  Difference between the ICIQ-SF score at the end of the pelvic floor rehablitation sessions and the ICIQ-SF score at 12 months and at 24 months in the control group
Urinary incontinence management 12 and 24 months after the end of the pelvic floor rehabilitation sessions in the intervention group | at 12 and 24 months
  New management of urinary incontinence, defined by new pelvic floor rehabilitation sessions, urinary incontinence or prolapse surgery, initiation of anticholinergic treatment, or any other therapy for urinary urinary at 12 and 24 months
Urinary incontinence management 12 and 24 months after the end of the pelvic floor rehabilitation sessions in the control group | at 12 and 24 months
  New management of urinary incontinence, defined by new pelvic floor rehabilitation sessions, urinary incontinence or prolapse surgery, initiation of anticholinergic treatment, or any other therapy for urinary urinary at 12 and 24 months
Impact of the videos on Knowledge and Satisfaction Ratings | after each video of the program, once a week for 4 weeks
  Difference in correct answers on questionnaires before and after each video, and satisfaction rating (0 to 10) after each video of the program
Usage of the videos provided in the intervention group | at the end of the video-based education program, 5 weeks after inclusion
  number of views for each video, time of day, total time spent on viewings (automatically collected via the connection platform)
Physical activity evolution after pelvic floor rehabilitation in the entire population and afetr 12 and 24 months | from inclusion to the end of the pelvic floor rehabilitation sessions (an average of 3 months), and after 12 and 24 months after the end of rehabilitation
  Compare the evolution of physical activity practice (intensity) from inclusion to the end of the pelvic floor rehabilitation sessions and after 12 and 24 months
Urinary incontinence score between the 2 groups according the UI type | at the end of the video-based education program versus the paper information document, 5 weeks after inclusion
  ICIQ-SF score at the end of the video-based education program vs the paper information document according to the UI type
Urinary incontinence score according to the dimensions of the Urinary Leakage Questionnaire | after the video-based education program, 5 weeks after inclusion
  to compare the ICIQ-SF score in each of the dimensions of the urinary leakage circumstances questionnaire after the video-based education program versus the paper information document

CONTACTS AND LOCATIONS:
Overall Officials: Anne Cecile Pizzoferrato, M.D, Study Director — University Hospital Center of Poitiers
Locations (12):
- France (12):
  - Mme ROSSIGNOL Marie - Kinésithérapeute - 5 place du Lavoir, Buxy
  - Mme BLANCHARD Véronique - Kinésithérapeute, Chanceaux-sur-Choisille
  - Mme GIRARD Delphine - kinésithérapeute - 14 rue de la Liberté, Embrun
  - Mme LIAGRE Blandine - Kinésithérapeute - 120 rue de Chanzy, Hellemmes-Lille
  - Mme BESSON Alice - Kinésithérapeute - 22 rue Benjamin Franklin, La Roche-sur-Yon
  - Mme OLIVIER Mathilde - Groupe médical du Barry - 34 Bis Rue du Quatre Septembre, Montignac
  - Mme CALONNE Hélène - Kinésithérapeute - 23 rue Franiatte, Montigny-lès-Metz
  - Mme LE TILLY Marine - Kinésithérapeute - 181 rue Legendre, Paris
  - Mme GIEN Isabelle - Kinésithérapeute - 2 Rue Adrienne Bolland, Saint-Jean-de-Braye
  - Mme LACOMBE Florence - Kinésithérapeute - 2 Rue Gabriel Durand, Saint-Médard-en-Jalles
  - Mme RIERE Claire - Kinésithérapeute - 62 Route de Saint-Aubin, Saint-Médard-en-Jalles
  - Mme GRUYER DROUET Laurence - Kinésithérapeute - 7 Rue Jean Baptiste Clément, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided